CLINICAL TRIAL: NCT07238764
Title: A Prospective Randomized Pilot Study of Early DAPT Discontinuation Based on Optical Coherence Tomography in High-Bleeding Risk Patients With Diabetes Mellitus Following Polymer-Free Amphilimus-Eluting Stent Implantation
Brief Title: OCT-based DAPT Cessation in HBR Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Conrady Alexandra, Deputy General Director for Research of the Almazov National Medical Research Center of the Ministry of Health of the Russian Federation, Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCT-DAPT
Record Dates: First submitted 2025-05-09; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: High Bleeding Risk Patients; DAPT(Dual Antiplatelet Therapy); Coronary Artery Disease; Diabetes Mellitus
Keywords: Optical coherence tomography; dual antiplatelet therapy; amphilimus-eluting stent; high-bleeding risk; diabetes mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard DAPT (6 months) (No Intervention): Standard DAPT therapy according to clinical guidelines
- Short DAPT (1 month) (Experimental): DAPT cessation at 1 month post-PCI based on optical coherence tomography results
  Interventions: Procedure: Optical Coherence Tomography-based early DAPT discontinuation

INTERVENTIONS:
Procedure: Optical Coherence Tomography-based early DAPT discontinuation — Within one month after the index PCI, participants in the short DAPT group underwent coronary angiography with OCT assessment of the implanted stents. If prespecified OCT criteria for adequate arterial healing were met (i.e., ≥80% neointimal strut coverage), DAPT was discontinued immediately, and SAPT with P2Y12 inhibitors was prescribed for up to six months.
  Arms: Short DAPT (1 month)

SUMMARY:
This study investigates whether patients with diabetes mellitus (DM) and a high risk of bleeding can safely stop dual antiplatelet therapy (DAPT) earlier than usual after receiving a special type of stent called a polymer-free amphilimus-eluting stent. DAPT, which combines aspirin and a P2Y12 inhibitor, is typically prescribed for six months after stent placement to prevent blood clots. However, in patients at high risk of bleeding, stopping DAPT early may be beneficial if the artery has healed properly.

The study uses optical coherence tomography (OCT), a high-resolution imaging tool, to assess how well the artery has healed after stent placement. If OCT shows that at least 80% of the stent is covered by new tissue after one month, patients in the short DAPT group stop taking DAPT and switch to a single antiplatelet drug for up to six months. In the standard DAPT group, patients continue taking both drugs for the full six months.

The goal of the study is to determine whether early DAPT discontinuation guided by OCT is as safe as the standard six-month treatment. The study focuses on two main outcomes: (1) how well the artery heals, measured by the percentage of stent coverage seen on OCT, and (2) the occurrence of major complications such as heart attack, stroke, or severe bleeding over 12 months.

This research is important because patients with diabetes often face delayed healing and a higher risk of blood clots, making it challenging to balance the risks of clotting and bleeding. The polymer-free amphilimus-eluting stent used in this study is designed to promote faster healing and reduce inflammation, potentially allowing for safer early DAPT discontinuation. Additionally, OCT provides precise information about arterial healing, helping doctors make personalized decisions about when to stop DAPT.

By comparing the safety and effectiveness of short DAPT versus standard DAPT, this study aims to improve treatment strategies for high-risk patients, reducing the risk of both bleeding and clot-related complications. If successful, this approach could lead to more tailored and safer antiplatelet therapy for patients with diabetes and high bleeding risk.

DETAILED DESCRIPTION:
This study investigates the safety and feasibility of early DAPT discontinuation guided by OCT findings in high-bleeding-risk patients with DM who undergo PCI with a polymer-free amphilimus-eluting stent. The research focuses on balancing the risks of bleeding and stent thrombosis, two critical complications associated with prolonged DAPT use, particularly in diabetic patients who are predisposed to delayed arterial healing and heightened thrombogenicity.

Study Design This is an investigator-initiated, single-center, prospective, randomized pilot trial designed to compare two DAPT strategies: short DAPT (OCT-guided discontinuation after 1 month) and standard DAPT (6 months). Eligible patients were randomized in a 1:1 ratio into the two groups, and all participants underwent PCI with the implantation of a polymer-free amphilimus-eluting stent (Cre-8, Alvimedica, Turkey). The study adheres to the principles of the Declaration of Helsinki and International Conference on Harmonization-Good Clinical Practice guidelines and was approved by the local ethics committee.

Patient Population The study included patients aged 18 years or older with known diabetes mellitus (type 1 or type 2), coronary artery disease (CAD) suitable for drug-eluting stent (DES) implantation, and a high-bleeding risk as defined by the Academic Research Consortium (ARC) or a Precise-DAPT score ≥ 25. Key exclusion criteria included acute coronary syndrome (ACS) or active bleeding at the time of randomization, severe renal impairment (glomerular filtration rate [GFR] ≤ 20 ml/min), and reduced left ventricular ejection fraction (LVEF ≤ 30%). A total of 40 patients were enrolled and randomized into the two study arms.

Interventions All participants received a loading dose of 300 mg of acetylsalicylic acid (ASA) and 600 mg of clopidogrel before PCI. The procedure was performed under local anesthesia with anticoagulation using unfractionated heparin (UFH) at a dose of 100 IU per kg. Full revascularization and adequate post-dilation were mandatory in both groups. In the short DAPT group, stent implantation was guided by OCT to ensure optimal stent strut apposition.

Within one month after PCI, patients in the short DAPT group underwent another OCT assessment to evaluate arterial healing. Early DAPT discontinuation was based on favorable OCT findings, defined as ≥80% neointimal strut coverage. OCT was performed using a commercially available system (Optis, Abbott, USA) and catheters (DragonFly Optis, Abbott, USA) according to a standardized protocol. Cross-sectional OCT images were analyzed at 2 mm intervals along the entire stented segment. For each analyzed segment, the total number of struts and uncovered struts (with no visible intimal coverage) were counted. Neointimal strut coverage was estimated as the total number of covered struts divided by the total number of analyzed struts.

If favorable OCT findings were observed, DAPT was discontinued, and single antiplatelet therapy (SAPT) with 75 mg of clopidogrel daily was prescribed for up to six months. In cases where OCT findings did not meet the predefined criteria, patients were switched to the standard DAPT regimen. In the standard DAPT group, patients continued dual antiplatelet therapy for the recommended duration of six months. After six months, all patients were transitioned to ASA only. Patients requiring oral anticoagulation were additionally prescribed non-vitamin K antagonist oral anticoagulants (NOACs) as per their clinical indications, alongside either DAPT or SAPT.

Endpoints The primary efficacy endpoint was the percentage of covered stent struts assessed by OCT at 1 month. This parameter was selected as a key marker of arterial healing, predictor of stent thrombosis risk, and indicator of safe DAPT abbreviation. The primary safety endpoint, defined as net adverse clinical events (NACE), included the incidence of cardiac death, non-fatal myocardial infarction (MI), stroke, or major bleeding (BARC types 2, 3, or 5). Secondary endpoints included the incidence of stent thrombosis and other major adverse cardiovascular events (MACE). Bleeding complications were assessed according to the Bleeding Academic Research Consortium (BARC) criteria.

Key Findings At 1 month, OCT analysis of 561 cross-sections in the short DAPT group showed a mean strut coverage of 87.4 ± 5.1%, with only one patient failing to meet the predefined coverage threshold (≥80% neointimal strut coverage) and subsequently transitioning to the standard DAPT regimen. During the 12-month follow-up period, no cardiac deaths, strokes, or stent thrombosis were reported in either group. Non-fatal non-target vessel myocardial infarctions occurred in one patient in each group. Major bleeding events were reported in three patients in the standard DAPT group and one patient in the short DAPT group. The cumulative incidence of NACE was numerically lower in the short DAPT group compared to the standard DAPT group (10% vs. 20%, p = 0.66), although the difference did not reach statistical significance.

Discussion This pilot study demonstrates the potential of OCT-guided early DAPT discontinuation in high-bleeding-risk patients with diabetes mellitus undergoing PCI with a polymer-free amphilimus-eluting stent. The favorable healing profile observed at 1 month suggests that this strategy may help balance the risks of bleeding and stent thrombosis. The absence of stent thrombosis and a numerically lower rate of major bleeding events in the short DAPT group align with emerging evidence supporting personalized DAPT strategies.

Recent landmark trials, such as MASTER-DAPT and STOPDAPT-2, have shown that short DAPT regimens in high-bleeding-risk populations are non-inferior to standard DAPT in terms of ischemic outcomes while significantly reducing bleeding events. These findings emphasize the importance of patient-centric decision-making in tailoring DAPT durations. The PROTECT-OCT registry and subsequent studies have highlighted the utility of OCT in assessing endothelial coverage and guiding early DAPT discontinuation. Our findings further support the role of OCT in identifying patients at low risk for stent thrombosis when DAPT is abbreviated.

The polymer-free amphilimus-eluting stent used in this study offers unique advantages, including a carbonized surface for improved hemocompatibility and an abluminal coating with long-chain fatty acids targeting inflammation and hyperproliferation. These attributes may enhance arterial healing, particularly in diabetic patients who are predisposed to delayed endothelialization.

Limitations As a single-center trial with a small sample size, the results should be interpreted with caution. While OCT is a promising tool for guiding DAPT strategies, its widespread implementation may be limited by cost and availability. Additionally, the 12-month follow-up period may not fully capture late adverse events, which are particularly relevant in high-risk populations.

Conclusion This pilot study demonstrates the feasibility and safety of OCT-guided early DAPT discontinuation in high-bleeding-risk patients with diabetes mellitus after polymer-free amphilimus-eluting stent implantation. The favorable healing profile observed at 1 month suggests the potential of this strategy to balance the risks of bleeding and stent thrombosis. However, larger multicenter trials are needed to validate these findings and further explore the role of OCT in tailoring antiplatelet therapy durations in high-risk populations.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (type 1 or type 2)
* Coronary artery disease (CAD) suitable for drug-eluting stent (DES) implantation
* High-bleeding risk as defined by the Academic Research Consortium (ARC) or a Precise-DAPT score ≥ 25

Exclusion Criteria:

* Acute coronary syndrome (ACS)
* Active bleeding at the time of randomization
* Known renal impairment (glomerular filtration rate [GFR] ≤ 20 ml/min)
* Reduced left ventricular ejection fraction (LVEF ≤ 30%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-12 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
The percentage of covered stent struts assessed by OCT at 1 month. The primary safety endpoint, defined as net adverse clinical events (NACE), included the incidence of cardiac death, non-fatal myocardial infarction (MI), stroke, or major bleeding. | 1 month

SECONDARY OUTCOMES:
Incidence of stent thrombosis and other MACE. Bleeding complications were assessed according to the BARC criteria. | The follow-up period was 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra O. Conradi, PhD, Study Chair — Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Locations (1):
- Almazov National Medical Research Center of the Ministry of Health of the Russian Federation, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No